CLINICAL TRIAL: NCT01783496
Title: Clinical Comparison of the Thermage CPT™ System's Framed and Pattern Tips for Treatment of Facial and Neck Laxity
Brief Title: Thermage CPT for Treatment of Facial and Neck Laxity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valeant Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-136-TM-T
Record Dates: First submitted 2013-01-31; First posted 2013-02-05 (Estimated); Results first posted 2014-11-17 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: Skin Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Framed Tip (Active Comparator): Treatment with Thermage CPT Framed Tip
  Interventions: Device: Thermage CPT
- Pattern Tip (Experimental): Treatment with the Thermage CPT Pattern Tip
  Interventions: Device: Thermage CPT
- Pattern Tip Group 2 (Experimental): Treatment with the Thermage CPT Pattern tip
  Interventions: Device: Thermage CPT
- Total Tip (Experimental): Treatment with the Thermage CPT Total tip
  Interventions: Device: Thermage CPT
- Framed and Patterned Tip (Experimental): Split face treatment with the Thermage CPT Framed and Patterned tips
  Interventions: Device: Thermage CPT
- Total and Patterned Tip (Experimental): Split face treatment with the Thermage CPT Total and Patterned tips
  Interventions: Device: Thermage CPT

INTERVENTIONS:
Device: Thermage CPT — Treatment with Thermage patterned, total, or framed tip

SUMMARY:
The purpose of this study to evaluate treatment with the Thermage CPT system for facial and neck laxity.

ELIGIBILITY:
Inclusion Criteria:

* 25 - 65 years of age
* Moderate facial and neck laxity
* Subject has the ability to follow the study instructions, is willing to be available on the specific required study visit days, and is willing to complete all study visit procedures and assessments.
* Subject must understand the research nature of this study and sign an Institutional Review Board (IRB)-approved informed consent prior to the performance of any study specific procedure or assessment.
* Subject agrees not to undergo excluded procedures on the face and neck for the duration of study.

Exclusion Criteria:

* Subject is pregnant or breast feeding, or trying to become pregnant for three months prior to or during the study.
* Pacemaker, internal defibrillator, or other implanted electronic device
* Subject has an active localized infection in the treatment area(s) or an uncontrolled systemic infection.
* Subject has had prior cosmetic procedures on the treatment area(s) within six months of the baseline visit.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Wheeland, MD, Principal Investigator
Locations (1):
- Solta Medical Aesthetic Center, Hayward, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Pattern Tip: Treatment with the Thermage CPT Pattern Tip Using Super-Pass Technique
- Pattern Tip Group 2: Treatment with the Thermage CPT Pattern tip Using Staggered-Pass Technique
Period: Overall Study
Arm/Group | Framed Tip | Pattern Tip | Pattern Tip Group 2 | Total Tip | Framed and Patterned Tip | Total and Patterned Tip
Started | 10 | 10 | 10 | 10 | 5 | 5
Completed | 9 | 10 | 10 | 8 | 5 | 4
Not Completed | 1 | 0 | 0 | 2 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Framed Tip | Pattern Tip | Pattern Tip Group 2 | Total Tip | Framed and Patterned Tip | Total and Patterned Tip | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 5 | 5 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (6.7) | 51.2 (8.1) | 49.1 (7.9) | 52.2 (7.5) | 51.0 (9.3) | 53.2 (8.0) | 51.6 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 6 | 10 | 2 | 5 | 42
  Male | 1 | 0 | 4 | 0 | 3 | 0 | 8
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 10 | 5 | 5 | 50
Mean Fasil Laxity Scale [Mean (Standard Deviation); unit: units on a scale] — (Fasil Laxity Scale: 0 = absent - 5 = severe)
  units on a scale | 2.7 (0.4) | 2.6 (0.5) | 2.7 (0.3) | 2.7 (0.8) | 2.5 (0.4) | 3.0 (0.5) | 2.7 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Laxity
Description: Improvement in facial and neck laxity 6 months following treatment as assessed by Study Investigator using a Quartile Improvement Scale score based upon a five point grading System: 4 - Very Significant Improvement (76-100%), 3 - Marked Improvement (51-75%), 2 - Moderate Improvement (26-50%), 1 - Minor/Mild Improvement (1-25%), or 0 - No Improvement.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Framed Tip | Pattern Tip | Pattern Tip Group 2 | Total Tip | Framed and Patterned Tip | Total and Patterned Tip
Number analyzed (Participants) | 9 | 10 | 10 | 8 | 5 | 4
units on a scale | 0.6 (0.5) | 1.0 (0.5) | 0.9 (0.5) | 1.3 (0.8) | 0.9 (0.3) | 1.4 (0.4)

2. Secondary Outcome: Improvement in Skin Laxity (Subject Self-assessed)
Description: Improvement in facial and neck laxity 6 months following treatment as self-assessed by subjects using a Quartile Improvement Scale score based upon a five point grading System: 4 - Very Significant Improvement (76-100%), 3 - Marked Improvement (51-75%), 2 - Moderate Improvement (26-50%), 1 - Minor/Mild Improvement (1-25%), or 0 - No Improvement.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Framed Tip | Pattern Tip | Pattern Tip Group 2 | Total Tip | Framed and Patterned Tip | Total and Patterned Tip
Number analyzed (Participants) | 9 | 10 | 10 | 8 | 5 | 4
units on a scale | 0.9 (0.9) | 1.4 (0.9) | 1.1 (0.5) | 1.2 (0.8) | 1.3 (1.1) | 2.4 (1.0)

3. Secondary Outcome: Subject Satisfaction With Treatment Results
Description: subjects were asked to provide satisfaction with treatment results, using the Likert Satisfaction Scale. Scoring was based upon a five point grading System: 5 - Very Satisfied, 4 - Satisfied, 3 - Neither Satisfied nor Dissatisfied, 2 - Dissatisfied, or 1 - Very Dissatisfied.
  Data are presented as the proportion of subjects showing improvement as defined as a score of 4 or greater ('satisfied' or 'very satisfied').
Time Frame: 6 months
Measure: Number; unit: percentage of subjects satisfied
Arm/Group | Framed Tip | Pattern Tip | Pattern Tip Group 2 | Total Tip | Framed and Patterned Tip | Total and Patterned Tip
Number analyzed (Participants) | 9 | 10 | 10 | 8 | 5 | 4
percentage of subjects satisfied | 56 | 60 | 80 | 38 | 60 | 75

ADVERSE EVENTS:
Arm/Group | Framed Tip | Pattern Tip | Pattern Tip Group 2 | Total Tip | Framed and Patterned Tip | Total and Patterned Tip
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/10 | 0/10 | 1/10 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 3/10 | 6/10 | 1/10 | 6/10 | 2/5 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Framed Tip (N=10) | Pattern Tip (N=10) | Pattern Tip Group 2 (N=10) | Total Tip (N=10) | Framed and Patterned Tip (N=5) | Total and Patterned Tip (N=5)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to treatment
Exploratory Vaginal Surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unrelated to treatment
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Framed Tip (N=10) | Pattern Tip (N=10) | Pattern Tip Group 2 (N=10) | Total Tip (N=10) | Framed and Patterned Tip (N=5) | Total and Patterned Tip (N=5)
Surface irregularity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intermittent itching (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Mild discomfort in treatment area (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jawline sensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cold (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to treatment
Tooth infection (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — Unrelated to treatment
Cellular atypia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Unrelated to treatment
Gout (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to treatment
Bruise due to fall (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to treatment
Erythema due to scratch (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated to treatment
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to treatment
hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to treatment
Pancreatitis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to treatment
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to treatment
Gum grafting (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to treatment
Rash due to sunscreen (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to treatment
Accidental injestion of marijuana (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unrelated to treatment
Seasonal allergies (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unrelated to treatment
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unrelated to treatment
Dental procedure (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unrelated to treatment
Hangnail infection (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unrelated to treatment
Sleep apnea (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unrelated to treatment
Hashimoto's disease (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unrelated to treatment
Vaginal bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unrelated to treatment
Headache (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unrelated to treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator shall notify Sponsor of the intent to publish or present independent Study Data, and agrees not to publish or publicly present and/or discuss such data, Investigator's current findings and/or the results of the Study independently without the express written consent of Sponsor, which consent may be withheld. Prior to submission for publication or presentation, all draft manuscripts must be submitted, reviewed and approved by Sponsor for confidential material.